Safety of TofAcitinib in Routine Care Patients With Rheumatoid Arthritis (STAR-RA) - Cardiovascular Endpoints

May 19, 2021

NCT04772248

## 1. Comparison Details

#### a. Intended aim(s)

- To compare the risk of cardiovascular events (including myocardial infarction or stroke), between patients treated with tofacitinib and patients treated with TNF inhibitors (TNFi) for rheumatoid arthritis (RA) among, 1) "real world evidence (RWE)" cohorts including routine care patient population from the US and, 2) "Randomized controlled trial (RCT) DUPLICATE" cohorts including routine care patient population who meet inclusion and exclusion criteria of the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis ("ORAL Surveillance", NCT02092467) clinical trial.
- To examine the risk of myocardial infarction, stroke, heart failure hospitalization, coronary revascularization, and all-cause mortality as separated endpoints when comparing tofacitinib with TNFi in patients with RA among, 1) "real world evidence (RWE)" cohort including routine care patient population from the US and, 2) "Randomized controlled trial (RCT) DUPLICATE" cohort including routine care patient population who meet inclusion and exclusion criteria of the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis ("ORAL Surveillance", NCT02092467) clinical trial.

### b. Primary endpoint

Major adverse cardiovascular events (MI and stroke)

## 2. Person responsible for implementation of analysis

Hemin Lee, MD, MPH will implement the study design and analysis in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps will be recorded and the implementation history will be archived in the platform. Propensity score (PS) fine stratification weighting will be implemented using SAS statistical software (SAS Institute, Cary, NC).

#### 3. Data Source(s)

US MarketScan, 2012-2018 Optum, 2012-2020 Medicare Claims Database, 2012-2017

## 4. Study Design Diagrams

### Figure 1. Inclusion and Exclusion Criteria for RWE and RCT Duplicate Cohorts

#### **Real World Evidence Cohorts**

#### **Inclusion Criteria**

- Patients treated with tofacitinib or TNF inhibitors in MarketScan (2012-2018), Optum (2012-2020), and Medicare fee-for-service (Parts A, B and D; 2012-2017)
- · At least 365 days of continuous enrollment in health plan prior to and including cohort entry date
- At least 2 RA codes between 7 and 365 days apart

#### **Exclusion Criteria**

- Index drug in 365 days prior to cohort entry date (prevalent users)
- < 18 years of age (Optum, MarketScan), < 65 (Medicare)</li>
- Missing data on age or gender
- Nursing home or hospice admission
- TNFi users with prior prescriptions of JAK inhibitors (tofacitinib, upadacitinib, or baricitinib)
- TNFi users initiating with multiple TNFi on same date
- Tofacitinib users with prior prescriptions of baricitinib, upadacitinib
- · Tofacitinib users initiating treatment with tofacitinib and baricitinib (or upadacitinib) on same day

#### **RCT-Duplicate Cohorts**

#### **Additional Inclusion Criteria**

- · Patients with at least one prescription of methotrexate
- Patients with at least one cardiovascular risk factor (including smoking, hypertension, dyslipidemia, diabetes mellitus, ischemic heart disease, family history of ischemic heart disease)

#### **Additional Exclusion Criteria**

- < 50 years of age (Optum, MarketScan), < 65 (Medicare)</p>
- · Patients recently hospitalized with infections
- · Pregnant patients

Figure 2: Study Design for RWE Cohorts



Figure 3: Study Design for RCT-Duplicate Cohorts



#### 5. Cohort Identification

## a. Cohort Summary

This study will employ an active comparator, new user observational cohort study design comparing initiators of tofacitinib to tumor necrosis factor inhibitors (infliximab, adalimumab, certolizumab pegol, etanercept, and golimumab). The patients will be required to have continuous enrollment in their health plan during the baseline period of 365 days before initiation of tofacitinib or TNFi (cohort entry date). Follow-up begins the day after drug initiation.

There will be two independent study populations:

- 1) Real-World Evidence (RWE) cohorts: This study population will reflect the patients diagnosed with RA who are routinely treated and managed in setting of clinical practice.
- 2) <u>RCT-duplicate cohorts</u>: This study population will emulate "the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis" clinical trial ("ORAL Surveillance", **NCT02092467**). The inclusion and exclusion criteria of this RCT will be applied to this study population.

### b. Inclusion and Exclusion Criteria Common to RWE and RCT-duplicate Cohorts

Cohort entry date:

• First TNFi or tofacitinib dispensation/administration date

Inclusion criteria:

- Patients treated with tofacitinib or TNF inhibitors in IBM MarketScan (2012-2018), Optum (2012-2020), and Medicare fee-for-service (Parts A, B and D; 2012-2017)
- A minimum of 365 days of continuous enrollment in health plan prior to (and including) the cohort entry date
- Two diagnosis codes for RA in any setting in 365 days baseline period (diagnosis codes between 7 and 365 days apart)

#### Exclusion criteria:

- Index drug in 365 days prior to cohort entry date (prevalent users)
- Missing data on age or gender
- Admission to nursing facility or hospice on or prior to cohort entry date (ever look-back)
- TNFi users with history of any Janus kinase (JAK) inhibitors (tofacitinib, upadacitinib, or baricitinib) (ever look-back period)
- TNFi users initiating with more than one TNFi on same date
- Tofacitinib users with a prescription of baricitinib, upadacitinib (ever look-back period)
- Tofacitinib users initiating treatment on multiple JAK inhibitors on same day (tofacitinib and baricitinib, tofacitinib and upadacitinib)

### c. Exclusion criteria specific to RWE cohorts

Patients less than 18 years of age (MarketScan and Optum) and 65 years of age (Medicare) at cohort entry

## d. Inclusion criteria specific to RCT-duplicate cohorts

- Patients with at least one methotrexate dispensation (six months look-back period)
- Patients with at least one cardiovascular risk factor (including smoking, hypertension, dyslipidemia, diabetes mellitus, ischemic heart disease, family history of ischemic heart disease) (one-year look-back period)

### e. Exclusion criteria specific to RCT-duplicate cohorts

- Patients less than 50 years of age (MarketScan and Optum) and 65 years of age (Medicare) at cohort entry
- Patients recently hospitalized with infections (30-day look-back period)
- Pregnant patients (one year look-back period)

# 6. Variables

# a. Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of tofacitinib

## **Comparator:**

Initiators of tofacitinib will be compared to initiators of TNFi (infliximab, adalimumab, certolizumab pegol, etanercept, and golimumab)

# b. Covariates (assessed during 365 day baseline period, unless otherwise specified):

| Demographics and Lifestyle Factors | |
|---|---|
| Age on the cohort entry date | Calendar year of cohort entry |
| Gender | Obesity |
| Race | Smoking |
| Rheumatoid arthritis related factors | |
| csDMARDs use (methotrexate, hydroxychloroquin | e, Number of distinct csDMARDs |
| leflunomide, sulfasalazine) | |
| Glucocorticoids use (365 day baseline, within 60 | Number of distinct bDMARDs |
| days of baseline, cumulative dose) | |
| CVD factors | |
| Atrial Fibrillation | Coronary Artery Disease |
| Type 2 Diabetes | Heart Failure |
| Stroke or transient ischemic attack | Hypertension |
| Hyperlipidemia | Peripheral vascular disease |
| Venous thromboembolism | |

| Comorbid conditions | |
|---|---|
| Cancer (except non-melanoma skin cancer) | Inflammatory bowel disease |
| Chronic liver disease | Psoriasis |
| Chronic kidney disease (stage 3+) | Combined comorbidity index |
| Chronic obstructive pulmonary disease | Frailty score |
| Comedication use | |
| Antidepressant drugs (including serotonin- | Antihypertensive drugs (including angiotensin |
| norepinephrine reuptake inhibitors, selective | II receptor blockers, angiotensin converting |
| serotonin reuptake inhibitors, tricyclic | enzyme inhibitors, beta blockers, calcium |
| antidepressants) | channel blockers, diuretics, nitrates) |
| Non-steroidal anti-inflammatory drugs | Lipid lowering drugs (Statins and non-statins) |
| Selective Cox-2 inhibitors | Anti-arrhythmic drugs |
| Opioids | Anticoagulants |
| COPD drugs (bronchodilators, inhaled | Antiplatelets (including acetylsalicylic acid) |
| corticosteroids) | |
| Other hormonal agents/HRT | Non-insulin diabetes medications |
| | Insulin |
| Markers for healthy behavior, frailty, healthcare use | |
| Number of C-reactive protein tests ordered | Echocardiogram |
| Number of serum creatinine tests ordered | Cardiac stress test |
| Number of lipid tests | Colonoscopy |
| Number of outpatient visits | Flu Shot |
| Number of primary care physician visits | Mammography |
| Number of rheumatologist visits | Pap smear |
| Number of emergency department visits | Pneumococcal vaccine |
| Number of hospitalizations (any, recent) | PSA test |
| Number of hospital days | Total distinct brand drugs used |
| Cardiologist visits | Total distinct generic drugs used |
| Electrocardiogram | Number of unique prescription medications |

# 7. Outcome variables and study follow-up:

- **<u>Primary outcome</u>**: Composite cardiovascular adverse events (myocardial infarction, stroke). Outcome will be defined by one inpatient claim.
- Secondary outcomes: Inpatients claims for myocardial infarction, stroke, heart failure hospitalization, coronary revascularization (including coronary artery bypass grafting and percutaneous coronary intervention), all-cause mortality

| Outcome | Codes | Care Setting | Position |
|---|---|---|---|
| Myocardial | ICD-9 DX: 410.** (except 410.*2) | Inpatient | Primary/ |
| infarction | | | Secondary |
| | ICD-10 DX: I21.0-I21.4, I22.* | | - |
| Stroke | ICD-9 DX: 430.**, 431.**, 433.*1, 434.** (excluding 434.x0), 436.** | Inpatient | Primary |
| | ICD-10 DX: I60.**, I61.*, I63.*** | | |
| Heart failure | <u>ICD-9 DX</u> : 398.91, 402.*1, 404.*1, 404.*3, 428.** | Inpatient | Primary |
| hospitalization | | | |
| | <u>ICD-10 DX</u> : I09.81, I11.0, I13.0, I13.2, I50.** | | |
| Coronary | <u>ICD-9 PX</u> : 00.66, 36.03-36.34, (except 36.04) | Inpatient | Any |
| revascularization | | | |
| | ICD-10 PX: 0210*, 0211*, 0212*, 0213*, 021K0Z5, 021K4Z5, 021L0Z5, | | |
| | 021L4Z5, 0270***, 0271***, 0272***, 0273***, 02C0*Z6, 02C2*Z6, | | |
| | 02C00ZZ, 02C03ZZ, 02C04ZZ, 02C10ZZ, 02C1*Z6, 02C13ZZ, 02C14ZZ, | | |
| | 02C20ZZ, 02C23ZZ, 02C24ZZ, 02C3*Z6, 02C30ZZ, 02C33ZZ, 02C34ZZ, | | |
| | 02QA0ZZ, 02QB0ZZ, 02QC0ZZ, 02QA3ZZ, 02QA4ZZ, 02QB3ZZ, | | |
| | 02QB4ZZ, 02QC3ZZ, 02QC4ZZ | | |
| | <u>CPT-4</u> : 33140, 33141, 33510-33536, 33545, 33572, 92920, 92921, | | |
| | 92924, 92925, 92928, 92929, 92933, 92934,92937, 92938, 92941, | | |
| | 92943, 92944, 92973, 92980, 92981, 92982, 92984, 92995, 92996 | | |

## Safety of TofAcitinib in Routine care patients with Rheumatoid Arthritis (STAR-RA)-Cardiovascular Endpoints Protocol

| All-cause | Inpatient (Optum |
|-----------|------------------|
| mortality | and MarketScan) |
| | Any setting |
| | (Medicare) |

## 8. Study Follow-up Period:

For the primary analysis, we will implement an <u>as-treated</u> exposure definition. Follow-up will start the day after initiation of tofacitinib and TNFi and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of enrollment in the database
- End of the study period
- Date of treatment switch or drug discontinuation, defined as the date of the last continuous treatment episode of the index drug plus a defined grace period (i.e., discontinuation defined after 60 days of no prescription refills for the index exposure after the days supply end for the most recent dispensing)
- Death

For secondary analysis, we will implement, an *intention-to-treat* exposure definition. Follow-up will start the day after initiation of tofacitinib and TNFi and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of enrollment in the database
- End of the study period
- Death
- 365 days after the cohort entry date

#### 9. Propensity score fine stratification analysis

We will use a propensity-score (PS)-based approach to account for measured confounding in this study.<sup>2</sup> The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., tofacitinib) conditional on baseline covariates using multivariable logistic regression constructed separately in each data source.<sup>3</sup> On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. We will trim non-overlapping regions of the propensity score distributions.<sup>3</sup> Subsequently, we will use PS fine stratification weighting to achieve covariate balance between treatment groups.<sup>4</sup> We will create 50 PS strata, based on the distribution of PS in tofacitinib-treated patients. A weight of one will be assigned to tofacitinib users and TNF inhibitor initiators will be weighted proportional to the distribution of tofacitinib initiators in the PS stratum into which they fell to achieve covariate balance (Nexposed in PS stratum i/ Ntotal) (Nreference in PS stratum i/Ntotal reference).<sup>4</sup> This weighting strategy estimates the average treatment effect on the treated (ATT).<sup>4</sup>

We will report multiple diagnostics for PS analysis in this protocol. First, the PS distribution overlap will be provided between two groups before weighting.<sup>4</sup> The balance in each individual covariate between two treatment groups will also be reported before and after weighting using standardized differences.<sup>5,6</sup> Distribution of PS weights will be assessed and truncation strategies will be considered if necessary.

### 10. Statistical analysis plans

Descriptive statistics, including frequencies and proportions for categorical variables and mean, median, standard deviation (SD), interquartile range (IQR), and range (minimum, maximum) for continuous variables, will be used to summarize baseline characteristics for each study cohort. Standardized differences will be used to compare characteristics before and after PS fine stratification weighting.<sup>5,6</sup> Crude incidence rates and corresponding 95% confidence intervals (CI) will be reported for each study outcome. The primary analysis will consist of Cox proportional hazards model weighted using PS fine stratification weights and using an *as-treated* exposure definition. This model will generate weighted hazard ratio and 95% confidence interval when comparing tofacitinib with TNFi. We will also report difference in rates when comparing tofacitinib with TNFi and corresponding 95% CI in the weighted population. Results will be reported independently for each database. Effect estimates will also be pooled across three databases using fixed effects model.

We will also report cumulative incidence and the corresponding 95% CI independently for all outcomes and each study group. Pre-specified subgroup analysis will be conducted based on age (≤65 and > 65), sex, and baseline cardiovascular disease (RWE cohorts only). Secondary analysis will be conducted by using an *intention-to-treat* exposure definition whereby patients will be censored 365 days after initiation of treatment with tofacitinib or TNF inhibitors. We will also conduct propensity score matching where each patient initiating tofacitinib will be matched with those initiating TNFi using nearest

neighbor greedy matching without replacement using a caliper of 0.025 on the natural scale of the PS (1:1 matching).<sup>3,7</sup> Standardized differences will be used to compare characteristics before and after matching. In addition, we will examine the risk of cardiovascular outcomes and all-cause mortality by stratifying by number of previous prescriptions of biological DMARDs (no previous prescriptions of bDMARDs vs ≥1 prescription of bDMARDs). Finally, sensitivity analyses will be conducted by restricting the TNFi comparator group to only adalimumab and etanercept users and by using herpes zoster as a positive control outcome.<sup>8</sup>

### 11. References

- 1. Lund JL, Richardson DB, Sturmer T. The active comparator, new user study design in pharmacoepidemiology: historical foundations and contemporary application. *Curr Epidemiol Rep.* 2015;2(4):221-228.
- 2. Rosenbaum PR RD. The central role of the propensity score in observational studies for causal effects. . *Biometrika*. 1983;70(1):41-55.
- 3. Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. *Multivariate Behav Res.* 2011;46(3):399-424.
- 4. Desai RJ, Franklin JM. Alternative approaches for confounding adjustment in observational studies using weighting based on the propensity score: a primer for practitioners. *BMJ*. 2019;367:l5657.
- 5. Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Stat Med.* 2014;33(10):1685-1699.
- 6. Austin PC. Using the Standardized Difference to Compare the Prevalence of a Binary Variable Between Two Groups in Observational Research. *Communications in Statistics Simulation and Computation*. 2008;38(6):1228-1234.
- 7. Austin PC. A comparison of 12 algorithms for matching on the propensity score. *Stat Med.* 2014;33(6):1057-1069.
- 8. Pawar A, R D, N G, et al. Risk of admission to hospital for serious infection after initiating tofacitinib versus biologic DMARDs in patients with rheumatoid arthritis: a multidatabase cohort study. *Lancet Rheumat*. 2020;2(2):e84-e98.